CLINICAL TRIAL: NCT06685666
Title: Effects of Elastic Band Exercises Added to the Warm-Up Program on Shooting Performance and Viscoelastic Properties of Upper Extremity Muscles in Youth Female Handball Players
Brief Title: Effects of Band Exercises Added to the Warm-Up on Shooting and Viscoelastic Properties of Muscles in Handball Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MarmaraU-AYDOGDU-OZCELİK001
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Healthy Athletes; Handball Players
Keywords: Handball player; Warm-Up Exercise; Elastic Band Exercise; Viscoelastic Proporties of Muscle; Shooting Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- traditional warm-up method specific to handball (Active Comparator): Traditional handball warm-up consists of dynamic and static warm-ups and passing and shooting drills.
  Interventions: Other: traditional warm-up method specific to handball
- elastic band exercises added to the traditional warm-up method specific to handbal (Experimental): Elastic band exercises added to the traditional handball warm-up consists of exercises for the upper extremity muscles that are active during the throw.
  Interventions: Other: elastic band exercises added to the traditional warm-up

INTERVENTIONS:
Other: traditional warm-up method specific to handball — The traditional warm-up program specific to handball consists of 6 basic sections: static stretching, aerobic work, dynamic mobility exercises, passes and crosses, shooting on goal and shooting according to position, and lasts 17 minutes in total.
  Arms: traditional warm-up method specific to handball
Other: elastic band exercises added to the traditional warm-up — The experimental group will be given elastic band exercises for 6 weeks after the static and dynamic exercises in the traditional warm-up and then continue with the warm-up with the ball. The exercise program was planned progressively. The exercises will be done in the first 3 weeks, 2 sets of 10 repetitions with a light resistance band. Then the exercises will be done in 3 sets of 10 repetitions with a medium resistance band. There are 8 band exercises in total.This exercise; Flexion and Extension Exercise in Diagonal Pattern, Internal and external rotation with the arm next to the body and the elbow in 90 degrees flexion, Internal and external rotation with the arm in 90 degrees abduction and the elbow in 90 degrees flexion, Scaption Exercise, Rowing, Biceps and Triceps (elbow flexion and extansion exercise), Wrist Flexors and Extensors (wrist flexion and extansion exercise).
  Arms: elastic band exercises added to the traditional warm-up method specific to handbal

SUMMARY:
Today's handball has become a fast and fluid handball that expects superior performance from athletes. The aim of handball is to put the ball into the opponent's goal, so one of the most important parameters of sports performance is shooting performance.

Studies show that warm-up programs have a positive effect on sports performance. Warm-up programs are used to prevent possible injuries and to increase sports performance by increasing temperature and flexibility in muscle and connective tissue. Warm-up programs may also cause changes in muscle viscoelastic properties and thus affect performance.

Recently, new approaches have begun to be used in warm-up programs. Some of these are warm-ups with a resistance tire, a medicine ball, and a weight vest. When the literature was examined, the effects of the warm-up program with resistance bands on adolescent handball players were generally examined in the lower extremity, but no study was found examining the effects on the upper extremity. For this reason, the study was designed to examine the effect of elastic band exercises applied to the upper extremity in addition to the traditional warm-up program on shooting performance in adolescent female handball players and the change in the viscoelastic properties of the upper extremity muscle groups.

30 female handball players with an age range of 12-18 years will participate in the research. Athletes will be divided into two equal groups as control and experimental groups in a controlled, randomized manner. The control group will be given a traditional warm-up program 6 days a week for 6 weeks. The experimental group will be given a traditional warm-up program under the same training conditions and additional elastic band exercises. In order to examine the effects of the warm-up programs to be applied in the chronic period, goal shooting, Modified Push Up test, Medicine Ball Throwing test, Upper Extremity Y Balance Test will be performed before training and at the 6th week and muscle viscoelastic properties will be evaluated. At the same time, in order to examine the acute effects, the goal shooting and muscle viscoelastic properties will be evaluated after the first warm-up training.The investigators hope that our study will help coaches and physiotherapists working in this field during the training process by ensuring the active use of a warm-up program with elastic bands in handball players.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years old
* Female Gender
* Participating in active training at least 3-4 times a week
* Athletes who volunteer to participate in the study
* Having a license in handball

Exclusion Criteria:

* People with orthopedic, neurological or congenital problems
* Athletes with chronic illnesses
* People with upper extremity surgery history within the last year
* People with cognitive problems
* People with problems that will prevent the application of tests
* Having had a sports injury that would affect upper extremity shooting performance within the last six months

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Goal Shot (Shot Accuracy) | before warm-up program
  In order to evaluate the shooting performance of the handball players, they will be asked to shoot at the designated areas of the goal. Four yellow target areas measuring 50 cm x 50 cm will be determined on the right-left, bottom and top corners of the handball goal. Athletes will be asked to take balls 11 m away from the goal and shoot at the goal from 9 meters. Each athlete will be asked to shoot at each of the four targets 7 times. The test will consist of a total of 35 shots (Van Den Tillaar and Ettema 2003) . In this study, the most commonly used techniques in previous studies and matches regarding the shot will be used, namely the basic shot with leaning step and the jump shot technique (Ion 2014).
Goal Shot (Shot Accuracy) | Immediately after the first warm-up program
  In order to evaluate the shooting performance of the handball players, they will be asked to shoot at the designated areas of the goal. Four yellow target areas measuring 50 cm x 50 cm will be determined on the right-left, bottom and top corners of the handball goal. Athletes will be asked to take balls 11 m away from the goal and shoot at the goal from 9 meters. Each athlete will be asked to shoot at each of the four targets 7 times. The test will consist of a total of 35 shots (Van Den Tillaar and Ettema 2003) . In this study, the most commonly used techniques in previous studies and matches regarding the shot will be used, namely the basic shot with leaning step and the jump shot technique (Ion 2014).
Goal Shot (Shot Accuracy) | six week later
  In order to evaluate the shooting performance of the handball players, they will be asked to shoot at the designated areas of the goal. Four yellow target areas measuring 50 cm x 50 cm will be determined on the right-left, bottom and top corners of the handball goal. Athletes will be asked to take balls 11 m away from the goal and shoot at the goal from 9 meters. Each athlete will be asked to shoot at each of the four targets 7 times. The test will consist of a total of 35 shots (Van Den Tillaar and Ettema 2003) . In this study, the most commonly used techniques in previous studies and matches regarding the shot will be used, namely the basic shot with leaning step and the jump shot technique (Ion 2014).
Analysis of Muscle-Tone Evaluation Using a Myotonometer | before warm-up program
  The MyotonPRO (myotonometer) device will be used to objectively evaluate the mechanical properties of the muscles (Viir, Virkus et al. 2007). In our study we will measure the tone (Hertz- Hz) value of the Deltoideus, Bicepss Brachii, Triceps Brachii, Flexor Carpi Radialis and Extensor Digitorium muscles. The athletes to be measured will first lie down in a supine position for 10 minutes and rest. Measurements will be made in the supine and prone positions of the individual from the dominant and non-dominant side. To determine the point where the measurement will be made, the athlete will be asked to perform an isometric contraction of the relevant muscle and the most swollen area of the muscle will be marked (Gavronski, Veraksitš et al. 2007).To minimize error in measurement, 3 measurements will be made from the same marked point and the average of the 3 values will be recorded.
Analysis of Muscle-Tone Evaluation Using a Myotonometer | Immediately after the first warm-up program
  The MyotonPRO (myotonometer) device will be used to objectively evaluate the mechanical properties of the muscles (Viir, Virkus et al. 2007). In our study we will measure the tone (Hertz- Hz) value of the Deltoideus, Bicepss Brachii, Triceps Brachii, Flexor Carpi Radialis and Extensor Digitorium muscles. The athletes to be measured will first lie down in a supine position for 10 minutes and rest. Measurements will be made in the supine and prone positions of the individual from the dominant and non-dominant side. To determine the point where the measurement will be made, the athlete will be asked to perform an isometric contraction of the relevant muscle and the most swollen area of the muscle will be marked (Gavronski, Veraksitš et al. 2007).To minimize error in measurement, 3 measurements will be made from the same marked point and the average of the 3 values will be recorded.
Analysis of Muscle-Tone Evaluation Using a Myotonometer | six week later
  The MyotonPRO (myotonometer) device will be used to objectively evaluate the mechanical properties of the muscles (Viir, Virkus et al. 2007). In our study we will measure the tone (Hertz- Hz) value of the Deltoideus, Bicepss Brachii, Triceps Brachii, Flexor Carpi Radialis and Extensor Digitorium muscles. The athletes to be measured will first lie down in a supine position for 10 minutes and rest. Measurements will be made in the supine and prone positions of the individual from the dominant and non-dominant side. To determine the point where the measurement will be made, the athlete will be asked to perform an isometric contraction of the relevant muscle and the most swollen area of the muscle will be marked (Gavronski, Veraksitš et al. 2007).To minimize error in measurement, 3 measurements will be made from the same marked point and the average of the 3 values will be recorded.
Analysis of Muscle Stiffness Evaluation Using a Myotonometer | before warm-up program
  The MyotonPRO (myotonometer) device will be used to objectively evaluate the mechanical properties of the muscles (Viir, Virkus et al. 2007). In our study we will measure the stiffness (Newton/meter- N/ m) value of the Deltoideus, Bicepss Brachii, Triceps Brachii, Flexor Carpi Radialis and Extensor Digitorium muscles. The athletes to be measured will first lie down in a supine position for 10 minutes and rest. Measurements will be made in the supine and prone positions of the individual from the dominant and non-dominant side. To determine the point where the measurement will be made, the athlete will be asked to perform an isometric contraction of the relevant muscle and the most swollen area of the muscle will be marked (Gavronski, Veraksitš et al. 2007).To minimize error in measurement, 3 measurements will be made from the same marked point and the average of the 3 values will be recorded.
Analysis of Muscle Stiffness Evaluation Using a Myotonometer | Immediately after the first warm-up program
  The MyotonPRO (myotonometer) device will be used to objectively evaluate the mechanical properties of the muscles (Viir, Virkus et al. 2007). In our study we will measure the stiffness (Newton/meter- N/ m) value of the Deltoideus, Bicepss Brachii, Triceps Brachii, Flexor Carpi Radialis and Extensor Digitorium muscles. The athletes to be measured will first lie down in a supine position for 10 minutes and rest. Measurements will be made in the supine and prone positions of the individual from the dominant and non-dominant side. To determine the point where the measurement will be made, the athlete will be asked to perform an isometric contraction of the relevant muscle and the most swollen area of the muscle will be marked (Gavronski, Veraksitš et al. 2007).To minimize error in measurement, 3 measurements will be made from the same marked point and the average of the 3 values will be recorded.
Analysis of Muscle Stiffness Evaluation Using a Myotonometer | six week later
  The MyotonPRO (myotonometer) device will be used to objectively evaluate the mechanical properties of the muscles (Viir, Virkus et al. 2007). In our study we will measure the stiffness (Newton/meter- N/ m) value of the Deltoideus, Bicepss Brachii, Triceps Brachii, Flexor Carpi Radialis and Extensor Digitorium muscles. The athletes to be measured will first lie down in a supine position for 10 minutes and rest. Measurements will be made in the supine and prone positions of the individual from the dominant and non-dominant side. To determine the point where the measurement will be made, the athlete will be asked to perform an isometric contraction of the relevant muscle and the most swollen area of the muscle will be marked (Gavronski, Veraksitš et al. 2007).To minimize error in measurement, 3 measurements will be made from the same marked point and the average of the 3 values will be recorded
Analysis of Muscle Elasticity Evaluation Using a Myotonometer | before warm-up program
  The MyotonPRO (myotonometer) device will be used to objectively evaluate the mechanical properties of the muscles (Viir, Virkus et al. 2007). In our study we will measure the elasticity value of the Deltoideus, Bicepss Brachii, Triceps Brachii, Flexor Carpi Radialis and Extensor Digitorium muscles. The athletes to be measured will first lie down in a supine position for 10 minutes and rest. Measurements will be made in the supine and prone positions of the individual from the dominant and non-dominant side. To determine the point where the measurement will be made, the athlete will be asked to perform an isometric contraction of the relevant muscle and the most swollen area of the muscle will be marked (Gavronski, Veraksitš et al. 2007).To minimize error in measurement, 3 measurements will be made from the same marked point and the average of the 3 values will be recorded.
Analysis of Muscle Elasticity Evaluation Using a Myotonometer | Immediately after the first warm-up program
  The MyotonPRO (myotonometer) device will be used to objectively evaluate the mechanical properties of the muscles (Viir, Virkus et al. 2007). In our study we will measure the elasticity value of the Deltoideus, Bicepss Brachii, Triceps Brachii, Flexor Carpi Radialis and Extensor Digitorium muscles. The athletes to be measured will first lie down in a supine position for 10 minutes and rest. Measurements will be made in the supine and prone positions of the individual from the dominant and non-dominant side. To determine the point where the measurement will be made, the athlete will be asked to perform an isometric contraction of the relevant muscle and the most swollen area of the muscle will be marked (Gavronski, Veraksitš et al. 2007).To minimize error in measurement, 3 measurements will be made from the same marked point and the average of the 3 values will be recorded.
Analysis of Muscle Elasticity Evaluation Using a Myotonometer | six week later
  The MyotonPRO (myotonometer) device will be used to objectively evaluate the mechanical properties of the muscles (Viir, Virkus et al. 2007). In our study we will measure the elasticity value of the Deltoideus, Bicepss Brachii, Triceps Brachii, Flexor Carpi Radialis and Extensor Digitorium muscles. The athletes to be measured will first lie down in a supine position for 10 minutes and rest. Measurements will be made in the supine and prone positions of the individual from the dominant and non-dominant side. To determine the point where the measurement will be made, the athlete will be asked to perform an isometric contraction of the relevant muscle and the most swollen area of the muscle will be marked (Gavronski, Veraksitš et al. 2007).To minimize error in measurement, 3 measurements will be made from the same marked point and the average of the 3 values will be recorded.

SECONDARY OUTCOMES:
Medicine Ball Throw Test | before warm-up program
  The athletes upper extremity explosive strength and open kinetic chain function will be evaluated with this test and the test is a valid and reliable test (Stockbrugger and Haennel 2001). The athletes will be asked to stand in front of a wall with their feet shoulder-width apart and holding a medicine ball with both hands. They will then be asked to throw the medicine ball forward while holding it at head-high level (Van den Tillaar and Marques 2013). A 3 kg medicine ball will be used for the adolescent group in this test. The test will be applied 3 times and the data will be averaged.
Medicine Ball Throw Test | six week later
  The athletes upper extremity explosive strength and open kinetic chain function will be evaluated with this test and the test is a valid and reliable test (Stockbrugger and Haennel 2001). The athletes will be asked to stand in front of a wall with their feet shoulder-width apart and holding a medicine ball with both hands. They will then be asked to throw the medicine ball forward while holding it at head-high level (Van den Tillaar and Marques 2013). A 3 kg medicine ball will be used for the adolescent group in this test. The test will be applied 3 times and the data will be averaged.
Upper Extremity Y Balance Test | before warm-up programme
  It will be applied for the purpose of evaluating the upper extremity dynamic balance. This test will be performed on a platform created in the medial, inferolateral and superolateral directions prepared on the ground (Bauer, Panzer et al. 2021). The lines in the inferolateral and superolateral directions are placed at an angle of 45° and the pipe in the medial direction is placed at an angle of 135° to the others. The test will be applied to the athletes separately for the dominant and non-dominant arms. Before the test, the application protocols of the test will be explained to all athletes and they will be asked to try it once. The test will start with the modified push-up position and one hand on the balance point and the other hand on the line in the medial direction.Athletes will be asked to reach the farthest point on the line in a stable stance (Kara, Büyükturan et al. 2022). 3 repetitions will be required for each direction (Westrick, Miller et al. 2012).
Upper Extremity Y Balance Test | six week later
  It will be applied for the purpose of evaluating the upper extremity dynamic balance. This test will be performed on a platform created in the medial, inferolateral and superolateral directions prepared on the ground (Bauer, Panzer et al. 2021). The lines in the inferolateral and superolateral directions are placed at an angle of 45° and the pipe in the medial direction is placed at an angle of 135° to the others. The test will be applied to the athletes separately for the dominant and non-dominant arms. Before the test, the application protocols of the test will be explained to all athletes and they will be asked to try it once. The test will start with the modified push-up position and one hand on the balance point and the other hand on the line in the medial direction.Athletes will be asked to reach the farthest point on the line in a stable stance (Kara, Büyükturan et al. 2022). 3 repetitions will be required for each direction (Westrick, Miller et al. 2012).
Modified Push Up Test | before warm-up program
  The Modified Push Up Test will be used to measure the upper extremity strength and endurance of athletes (Hashim and Madon 2012). The athlete will be positioned on the mat with the knees and elbows in flexion position. The athlete will then be asked to push the upper body upwards by extending the elbows (Kara, Büyükturan et al. 2022). The number of correct movements within a 30-second period will be recorded.
Modified Push Up Test | six week later
  The Modified Push Up Test will be used to measure the upper extremity strength and endurance of athletes (Hashim and Madon 2012). The athlete will be positioned on the mat with the knees and elbows in flexion position. The athlete will then be asked to push the upper body upwards by extending the elbows (Kara, Büyükturan et al. 2022). The number of correct movements within a 30-second period will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Westrick RB, Miller JM, Carow SD, Gerber JP. Exploration of the y-balance test for assessment of upper quarter closed kinetic chain performance. Int J Sports Phys Ther. 2012 Apr;7(2):139-47. PMID 22530188
- [Background] Bauer J, Panzer S, Muehlbauer T. Side differences of upper quarter Y balance test performance in sub-elite young male and female handball players with different ages. BMC Sports Sci Med Rehabil. 2021 Nov 1;13(1):141. doi: 10.1186/s13102-021-00364-3. PMID 34724988
- [Background] van den Tillaar R, Marques MC. Reliability of seated and standing throwing velocity using differently weighted medicine balls. J Strength Cond Res. 2013 May;27(5):1234-8. doi: 10.1519/JSC.0b013e3182654a09. PMID 22744301
- [Background] Stockbrugger BA, Haennel RG. Validity and reliability of a medicine ball explosive power test. J Strength Cond Res. 2001 Nov;15(4):431-8. PMID 11726253
- [Background] Gavronski G, Veraksits A, Vasar E, Maaroos J. Evaluation of viscoelastic parameters of the skeletal muscles in junior triathletes. Physiol Meas. 2007 Jun;28(6):625-37. doi: 10.1088/0967-3334/28/6/002. Epub 2007 May 3. PMID 17664617
- [Background] van den Tillaar R, Ettema G. Instructions emphasizing velocity, accuracy, or both in performance and kinematics of overarm throwing by experienced team handball players. Percept Mot Skills. 2003 Dec;97(3 Pt 1):731-42. doi: 10.2466/pms.2003.97.3.731. PMID 14738333